CLINICAL TRIAL: NCT03595137
Title: The Effect of Simple Needle Guide Device for Ultrasound-guided Internal Jugular Vein Catheterization in Surgical Patients: a Randomized-controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1-2018-0027
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Patients Undergoing Surgery

STUDY DESIGN:
Intervention Model Description: 1. sono with simple needle guide device group
  2. sono only group
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sono with simple needle guide device group (Group D) (Experimental): sono with simple needle guide device Simple needle guide device was attached to the sono probe. Device was designed to assist the detection of the puncture site. After induction of anesthesia, sono-guided internal jugular vein cannulation was performed.
  Interventions: Device: Sono with Device
- sono only group (Group S) (Placebo Comparator): sono only group After induction of anesthesia, sono-guided internal jugular vein cannulation was performed.
  Interventions: Device: Sono only

INTERVENTIONS:
Device: Sono with Device — In Group D, simple needle guide device was attached to the sono probe. Device was designed to assist the detection of the puncture site. After induction of anesthesia, sono-guided internal jugular vein cannulation was performed.
  Arms: sono with simple needle guide device group (Group D)
Device: Sono only — In group S, sono-guided internal jugular vein cannulation was performed after induction of anesthesia
  Arms: sono only group (Group S)

SUMMARY:
The purpose of this study is to evaluate the effect of simple needle guide device for ultrasound-guided internal jugular vein catheterization in surgical patients

ELIGIBILITY:
Inclusion Criteria:

1. adult ( ≧19 years old)
2. patients undergoing elective surgery

Exclusion Criteria:

1. emergency surgery
2. patients under cervical immobilization
3. anatomical abnormality for Right internal jugular vein catheterization
4. infection or hematoma at puncture site
5. patients who did not need internal jugular vein catheterization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
First access success rate | up to 5 minutes after insertion of puncture needle
  First access success rate was defined as the number of sono-guided catheterization obtained within first attempt

SECONDARY OUTCOMES:
insertion time | 10 minutes after the beginning of the procedure
  defined as the time in seconds between the beginning of the procedure and guide-wire insertion
complication rate | 24 hours after surgery
  incidence of Pneumothorax, Haemothorax, Hydrothorax, carotid artery puncture, Hematoma, Malpositions, puncture of posterior wall of internal jugular vein
ease of procedure | 10 minutes after the beginning of the procedure
  In order to measure the degree of difficulty felt by the subjects during the procedure, a 100mm visual analogue scale was used to measure 10 difficulty levels (100mm; ease, 0mm ; difficult)
the number of separate skin puncture | 10 minutes after the beginning of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No